CLINICAL TRIAL: NCT04423094
Title: Foci of Tumor Heterogeneity in IDH1-mutated Diffuse Low-Grade Gliomas Reveal STAT3 Activation and Downregulation of the Phosphoethanolamine Enzyme ETNPPL Acting as a Negative Regulator of Glioma Growth
Brief Title: Foci of Tumor Heterogeneity in Diffuse Low-Grade Gliomas
Acronym: FDLGG
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0469
Record Dates: First submitted 2019-11-25; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Diffuse low-grade gliomas (DLGG) are slow-growing primary-cancer of the brain and spinal cord. They represent up to 15% of the developing tumors in those organs with fatal outcome for the patients because of their evolution. The reasons for this transformation towards more malignant tumors still remain ill defined. Previously, the research team in neuro oncology at Montpellier University Hospital found foci of tumor heterogeneity within 20 to 30 % of the patients developing a DLGG and published their results. The investigators assumed that those foci represent the early beginning of the transformation from a diffuse low-grade glioma to a glioblastoma, tumor with highly malignant cells and a life expectancy of two years in average for the patient.

Methods:

The investigators selected adult patients with no prior surgery nor neuro oncology treatment when enrolled. They presented a specific mutation for an enzyme of the metabolism named IDH1, standing for Isocitrate Dehydrogenase 1, found in 70% of DLGG. Patients were also selected because they presented foci of tumor heterogeneity. After obtaining their consent, the investigators studied by immunohistochemistry the pathways deregulated between the DLGG and the foci. The investigators also extracted RNAs, molecules expressing the life and metabolism of tumor cells, and compared them to know what genes were differentially expressed between the DLGG and the foci. All RNAs were tested for quality control prior to be processed further. The investigators then studied 8 patients with compliance with ethics, authorizations and institutional guidelines. Genes of interest were studied in vitro to assess their functions. The investigators found a barely described enzyme of the catabolism of the phosphoethanolamines and discovered a new anti-proliferative tumor-role for it.

•Discussion: The investigators first showed that foci have a higher percentage of p-STAT3+ cells which indicates STAT3 pathway activation in these cells. Phosphorylated STAT3 translocates to the cell nucleus to regulate many genes involved in proliferation, apoptosis and angiogenesis. As such, phosphorylation of STAT proteins, notably STAT3, is involved in the pathogenesis of many cancers, including GBM, by promoting cell cycle progression, stimulating angiogenesis, and impairing tumor immune surveillance.

The investigators found that ETNPPL RNA and protein are reduced in foci cells and absent in glioblastomas. This is consistent with glioma database analyses showing that ETNPLL expression is inversely correlated to STAT3 and MKI67 whose expression are higher in foci and glioblastomas. In addition, Kaplan-Meier analysis shows that patients with low expression of ETNPPL have lower overall survival These observations suggested that this enzyme may oppose glioma cells proliferation. The investigators demonstrated this hypothesis by overexpressing ETNPPL in 3 glioblastoma cell cultures. Two were sensitive to ETNPPL overexpression which reduced their growth while no effect was detected in Gli4 cells. These glioblastoma-derived cultures have different types of mutations.

DETAILED DESCRIPTION:
IDH1-mutated gliomas are slow-growing brain tumors which progress into high-grade gliomas. The early molecular events causing this progression are ill-defined. Previous studies revealed that 20% of these tumors already have transformation foci. These foci offer opportunities to better understand malignant progression. The investigators used immunohistochemistry and high throughput RNA profiling to characterize foci cells. These have higher p-STAT3 staining revealing activation of JAK/STAT signaling. They downregulate genes involved in Hippo/Yap pathway (AMOT, CCDC80, LIX1), Wnt signaling (CPE, DAAM2, GPR37, SFRP2), EGFR signaling (EPS15, MLC1), cytoskeleton and cell-cell communication (EZR, GJA1) while increasing SKA3, a kinetochore-associated protein. In addition, foci cells show reduced levels of the lipid metabolic ethanolamine-phosphate phospho-lyase (ETNPPL/AGXT2L1). This enzyme is involved in the catabolism of phosphoethanolamine involved in membrane synthesis. The investigators detected ETNPPL protein in glioma cells as well as in astrocytes in the human brain. Its nuclear localization suggests additional roles for this enzyme. ETNPPL expression is inversely correlated to glioma grade and the investigators found no ETNPPL protein in glioblastomas.

Overexpression of ETNPPL reduces the growth of glioma stem cells indicating that this enzyme opposes gliomagenesis. Collectively, these results suggest that a combined alteration in membrane lipid metabolism and STAT3 pathway promotes IDH1-mutated glioma malignant progression.

Tumors with foci of at least four millimeters in diameter, assessed by hematoxylin & eosin stainings, were selected. Four drills (two in foci and two in the other part of the tumor ) were performed in the FFPE tumor blocks using a two millimetres punch from a Tissue Micro Array apparatus in RNAse-free conditions. After the punches, the adequate selection of tumor areas was checked by hematoxylin & eosin stainings of sections. Total RNA was extracted using the Qiagen RNeasy FFPE kit, quantified with Nanodrop 1000 (Thermo Fisher) and the RNA integrity number (RIN) was determined using a Bioanalyzer 2100. The RIN was on average 2.5 but were still suitable for labelling and hybridization on DNA chips according to the Affymetrix technical department. After amplification and labelling with an Affymetrix WT Pico Kit, cDNA were hybridized on Human Gene 2.1 ST chips. Data were normalized with the Affymetrix Expression Console software (GC-RMA algorithm) and the RNA profiles were generated using the Affymetrix Transcriptome Analysis Console (3.1.0.5) software. Differentially expressed genes were selected on the basis of a linear fold change ≥ 1.1 and p-value ≤ 0.05 (n=8 tumors). The data that support the findings of our study are openly available at the functional genomics data Gene Expression Omnibus.

ELIGIBILITY:
Inclusion criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged between 18 and 70 years.
* Suffering from IDH1-mutated diffuse low-grade glioma.
* No pre operative nor oncology treatment prior to join the study.
* Signed informed consent form.

Exclusion criteria:

* Subject unable to read or/and write
* Grade 3 or 4 gliomas
* Tumor with IDH1-WT status

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An individual must fulfill all of the following criteria in order to be eligible for study enrollment Aged between 18 and 70 years, Suffering from IDH1-mutated diffuse low-grade glioma, No pre operative nor oncology treatment prior to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
statistically significant increase in the number of tumor cells | 1 day
  statistically significant increase in the number of tumor cells

SECONDARY OUTCOMES:
determine predictive markers of this tumor development | 1 day
  determine predictive markers of this tumor development

CONTACTS AND LOCATIONS:
Overall Officials: VALERIE RIGAUX, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC